CLINICAL TRIAL: NCT06573788
Title: Multidisciplinary Prehabilitation Management Pathway and Network Platform Construction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, ZIJIA LIU, associate chief physician, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ZJL-005
Record Dates: First submitted 2024-08-16; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer; Prehabilitation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Block randomized number will be prepared in advance and be hidden in the envelope. At the time of collecting the participants' baseline information, neither the participants nor the investigator knew which intervention the patients would receive. After the information was collected, the envelopes were opened to determine whether participants were assigned to the intervention or control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet+wearble device prehabilitation model (Experimental): Pre-rehabilitation components include smoking cessation, aerobic training, anaerobic exercise, nutritional optimization and psychological support.
  "Internet+" group using online application + wearable device management model
  Interventions: Behavioral: Internet + wearble device multimodal prehabilitation
- traditional prehabilitation model (Active Comparator): The traditional prehabilitation group used the traditional management model of preoperative education + paper records + regular weekly reminders from healthcare professionals
  Interventions: Behavioral: traditional multimodal prehabilitation

INTERVENTIONS:
Behavioral: Internet + wearble device multimodal prehabilitation — Use the Prehabilitation Learning Platform to learn what to do and follow along with the videos for follow up exercises
  Arms: Internet+wearble device prehabilitation model
Behavioral: traditional multimodal prehabilitation — The researchers used a prehabilitation manual to explain to subjects what they needed to do, and the patients went home and practiced on their own, recording the exercises daily
  Arms: traditional prehabilitation model

SUMMARY:
The goal of this clinical trial is to learn if "Prehabilitation model for Internet+ devices"improve patients' preoperative status and reduce the postoperative recovery time, postoperative complications，comparing to trditional prehabilitation model. The main questions it aims to answer are:

1. Does the Prehabilitation model for Internet+ devices works out?
2. Does"Prehabilitation model for Internet+ devices" better increase the patient's six-minute walk test distance?

Participants will:

Take Internet+devices model or traditional model to prehabilitation for 2-4weeks.

Test 6MWT before operation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years;
2. adults with suspected lung cancer proposed for VATS lobectomy/sublobar resection.

Exclusion Criteria:

1. Patient refusal;
2. ASA classification IV or higher;
3. Pre-neoadjuvant chemotherapy;
4. Inability to cooperate (psychiatric abnormalities, impaired consciousness, mental retardation);
5. Comorbidities cannot tolerate home rehabilitation or functional motor examination;
6. Inability to use a smartphone or read Chinese;
7. Average weekly moderate-intensity/high-intensity exercise of >90min/>60min.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
6 minute walking test distance, 6MWD | About 2-4 month before surgery(When deciding on surgery), 1 day before surgery, 30 days after surgery
  Using 6MWD as the primary assessment of patients' perioperative functional status and the primary endpoint of the study, patients were evaluated at enrollment, before surgery, and 30 days after surgery, respectively.

SECONDARY OUTCOMES:
Length of hospitalization | About 2-4 month before surgery(When deciding on surgery), 1 day before surgery, 30 days after surgery
postoperative complication | 30 days after surgery
pulmonary function | About 2-4 month before surgery(When deciding on surgery), 1 day before surgery, 30 days after surgery
  FVC
pulmonary function | About 2-4 month before surgery(When deciding on surgery), 1 day before surgery, 30 days after surgery
  FEV1
pulmonary function | About 2-4 month before surgery(When deciding on surgery), 1 day before surgery, 30 days after surgery
  FEV1/FVC
pulmonary function | About 2-4 month before surgery(When deciding on surgery), 1 day before surgery, 30 days after surgery
  MVV
grip | About 2-4 month before surgery(When deciding on surgery), 1 day before surgery, 30 days after surgery
  Using grip dynamometer to measure the grip strength of the patient's hand, measured in kg
NRS2002 Nutritional Risk Screening | About 2-4 month before surgery(When deciding on surgery), 1 day before surgery, 30 days after surgery
Hospital Anxiety and Depression Scale（HADS） | About 2-4 month before surgery(When deciding on surgery), 1 day before surgery, 30 days after surgery
  There are 14 questions in total, with four options for each question ranging from 0 to 3；0 to 7 indicating no symptoms, 8 to 10 indicating suspected anxiety or depression symptoms, and 11 to 21 indicating certain symptoms
Quality of Recovery-15（QOR-15） | About 2-4 month before surgery(When deciding on surgery), 1 day before surgery, 30 days after surgery
  A total of 15 questions, each question have 0-10 points, the higher the score means the better the recovery effect
World Health Organization Disability Assessment Schedule 2.0（WHODAS 2.0） | About 2-4 month before surgery(When deciding on surgery), 1 day before surgery, 30 days after surgery
  Questions are on a scale of 1-5, with a lower score indicating that the patient is generally better.

CONTACTS AND LOCATIONS:
Overall Officials: Zijia Liu, Principal Investigator — Peking Union Medical College Hospital

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT06573788/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT06573788/ICF_001.pdf